CLINICAL TRIAL: NCT05904054
Title: An Open-label and Single-center Phase IIa Trial to Evaluate the Immunogenicity and Safety of SARS-CoV-2 DNA Vaccine (ICCOV) in Healthy Subjects Aged 18-75 Years
Brief Title: Immunogenicity and Safety Study of SARS-CoV-2 DNA Vaccine (ICCOV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immuno Cure 3 Limited (Industry)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor
Organization: Immuno Cure Holding (HK) Limited (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICCOV_HK202301
Record Dates: First submitted 2023-06-02; First posted 2023-06-15 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
Keywords: ICCOV; COVID-19; DNA Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Adult-CoronaVac® group (Experimental): Aged 18-59 AND received 2 to 4 homologous doses of CoronaVac® at least 3 months prior to enrollment AND without SARS-CoV-2 infection history.
  Interventions: Biological: SARS-CoV-2 DNA Vaccine (ICCOV)
- Adult-Comirnaty® group (Experimental): Aged 18-59 AND received 2 to 4 homologous doses of Comirnaty® at least 3 months prior to enrollment AND without SARS-CoV-2 infection history.
  Interventions: Biological: SARS-CoV-2 DNA Vaccine (ICCOV)
- Adult-mixed group (Experimental): Aged 18-59 AND received 2 to 4 heterologous doses of CoronaVac® and Comirnaty® at least 3 months prior to enrollment AND without SARS-CoV-2 infection history; OR Aged 18-59 AND received 2 to 4 heterologous doses of CoronaVac® and Comirnaty® at least 3 months prior to enrollment AND recovered from SARS-CoV-2 infection at least 3 months prior to enrollment; OR Aged 18-59 AND received 2 to 4 homologous doses of CoronaVac® or Comirnaty® at least 3 months prior to enrollment AND recovered from SARS-CoV-2 infection at least 3 months prior to enrollment.
  Interventions: Biological: SARS-CoV-2 DNA Vaccine (ICCOV)
- Elderly-mixed group (Experimental): Aged 60-75 AND received 2 to 4 heterologous doses of CoronaVac® and Comirnaty® at least 3 months prior to enrollment AND without SARS-CoV-2 infection history; OR Aged 60-75 AND received 2 to 4 heterologous doses of CoronaVac® and Comirnaty® at least 3 months prior to enrollment AND recovered from SARS-CoV-2 infection at least 3 months prior to enrollment; OR Aged 60-75 AND received 2 to 4 homologous doses of CoronaVac® or Comirnaty® at least 3 months prior to enrollment AND without SARS-CoV-2 infection history; OR Aged 60-75 AND received 2 to 4 homologous doses of CoronaVac® or Comirnaty® at least 3 months prior to enrollment AND recovered from SARS-CoV-2 infection at least 3 months prior to enrollment.
  Interventions: Biological: SARS-CoV-2 DNA Vaccine (ICCOV)

INTERVENTIONS:
Biological: SARS-CoV-2 DNA Vaccine (ICCOV) — The SARS-CoV-2 DNA Vaccine (ICCOV) was developed by Immuno Cure Holding (HK) Limited.The product is a pre-filled syringe or a vial with an extractable volume of 0.5 mL. The unit dose strength is 1 mg/0.5 mL and the dose volume is 1.0 mL/dose.
  Other Names: ICCOV

SUMMARY:
This is an open-labeled, no placebo, Phase IIa clinical trial. The purpose of this study is to evaluate the immunogenicity and safety of one booster vaccine dose of SARS-CoV-2 DNA Vaccine (ICCOV) in adults aged 18 to 75 years who have received two to four dosese of COVID-19 vaccine.

DETAILED DESCRIPTION:
This is an open-labeled, no placebo, Phase IIa clinical trial to evaluate the immunogenicity and safety of one booster vaccine dose of SARS-CoV-2 DNA Vaccine (ICCOV) in adults aged 18 to 75 years who have received two to four dosese of COVID-19 vaccine. The primary purpose of this study is to evaluate cross-reactive T cell responses against SARS-CoV-2 prototype and epidemic variants induced by one booster dose of ICCOV. The secondary purposes are 1) to evaluate other variables of cross-reactive T cell responses against SARS-CoV-2 prototype and epidemic variants induced by one booster dose of ICCOV; 2) to evaluate humoral immunity responses against SARS-CoV-2 prototype and epidemic variants induced by one boosterdose of ICCOV; and 3) to evaluate the safety and reactogenicity of ICCOV.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to comply with all study requirements.
2. Give informed consent and sign informed consent form (ICF). For subjects who are unable to read or write, the consent must be witnessed by a literate third party not involved in the study.
3. BMI in between 18.5 and 30.0 kg/m2 (including upper and lower limits).
4. For each group, meet the following criteria regarding age, COVID-19 vaccination history (as confirmed by COVID-19 vaccination records), and SARS-CoV-2 infection history (as confirmed by the investigator according to WHO definitions, Appendix III):

   Group 1: Adult-CoronaVac® group

   - Aged 18-59 AND received 2 to 4 homologous doses of CoronaVac® at least 3 months prior to enrollment AND without SARS-CoV-2 infection history.

   Group 2: Adult-Comirnaty® group

   - Aged 18-59 AND received 2 to 4 heterologous doses of CoronaVac® and Comirnaty® at least 3 months prior to enrollment AND without SARS-CoV-2 infection history; OR

   Group 3: Adult-mixed group
   * Aged 18-59 AND received 2 to 4 heterologous doses of CoronaVac® and Comirnaty® at least 3 months prior to enrollment AND without SARS-CoV-2 infection history; OR
   * Aged 18-59 AND received 2 to 4 heterologous doses of CoronaVac® and Comirnaty® at least 3 months prior to enrollment AND recovered from SARS-CoV-2 infection at least 3 months prior to enrollment; OR
   * Aged 18-59 AND received 2 to 4 homologous doses of CoronaVac® or Comirnaty® at least 3 months prior to enrollment AND recovered from SARS-CoV-2 infection at least 3 months prior to enrollment.

   Group 4: Elderly-mixed group
   * Aged 60-75 AND received 2 to 4 heterologous doses of CoronaVac® and Comirnaty® at least 3 months prior to enrollment AND without SARS-CoV-2 infection history; OR
   * Aged 60-75 AND received 2 to 4 heterologous doses of CoronaVac® and Comirnaty® at least 3 months prior to enrollment AND recovered from SARS-CoV-2 infection at least 3 months prior to enrollment; OR
   * Aged 60-75 AND received 2 to 4 homologous doses of CoronaVac® or Comirnaty® at least 3 months prior to enrollment AND without SARS-CoV-2 infection history; OR
   * Aged 60-75 AND received 2 to 4 homologous doses of CoronaVac® or Comirnaty® at least 3 months prior to enrollment AND recovered from SARS-CoV-2 infection at least 3 months prior to enrollment.
5. Healthy subjects, or subjects with stable medical condition who have a pre-existing medical condition that does not meet any exclusion criteria. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months prior to enrollment.
6. Female subjects of childbearing potential with have negative pregnancy test shall be willing to practice continuous effective contraception and not to breastfeed until 12 months after ICCOV administration.

   * Nonchildbearing potential is defined as surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, hysterectomy) or postmenopausal. A follicle-stimulating hormone (FSH) level and the amenorrhea duration (e.g., amenorrhea for ≥ 12 consecutive months prior to screening without an alternative medical cause) may be measured at the discretion of the investigator to confirm postmenopausal status.
   * The effective contraceptive methods include sexual abstinence or adequate contraceptive measures such as intrauterine or implanted contraceptive device, oral contraceptives, injected or implanted contraceptives, sustained-release topical contraceptives, condoms (male), diaphragm, and cervical cap, etc.
7. Male subjects who are involved in heterosexual sexual activity must agree to practice adequate contraception (as described above) and refrain from donating sperm until 12 months after ICCOV administration.
8. Agreement to avoid blood donation during the study.

Exclusion Criteria:

1. Laboratory confirmed SARS-CoV-2 infection, defined by RT-PCR test.
2. Fever (oral temperature ≥ 37.5°C/axillary temperature ≥ 37.3°C) on the day of vaccination or within recent 72 hours.
3. Medical history of severe acute respiratory syndrome (SARS), middle east respiratory syndrome (MERS) within 12 months, and COVID-19 within 3 months prior to enrollment.
4. Abnormal laboratory tests of clinical significance involving hematology, serum biochemistry, coagulation function, or urinalysis as determined by the investigator.
5. Females who are pregnant or breastfeeding or those who plan to give birth in coming 12 months (including in female subjects or the female partners of male subjects).
6. Participated in other clinical trials and received any other investigational products within 1 month (or 5 half-lives of the drug, whichever is longer) prior to enrollment or plan to receive any other investigational products during the study.
7. History of severe allergies to any vaccine or drug, such as urticaria, dyspnea, edema, abdominal pain and other symptoms after administration, especially hypersensitivity to the components of ICCOV.
8. Have malignant tumor (except for skin basal cell carcinoma or carcinoma uterine cervix in situ) and immune disease (e.g., human immunodeficiency virus [HIV] infection, systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy, severe combined immunodeficiency disorder [SCID], and other immune disease that may influence immune response at the investigator's discretion).
9. Have other severe and/or uncontrolled conditions, including but not limited to, acute infectious disease, cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, hematology disease, endocrine disorder, psychiatric condition and neurological illness (e.g., Guillain-Barre Syndrome, uncontrolled epilepsy, etc.). Mild/moderate well-controlled comorbidities are allowed to participate as deemed appropriate by the investigator.
10. Received any investigational or licensed COVID-19 vaccine other than described in inclusion criteria, or any investigational or approved vaccine against a coronavirus (including but not limited to SARS-CoV-1 and MERS-CoV) at any time prior to enrollment.
11. Received any investigational or approved vaccines within 3 months prior to enrollment or plan to receive any other vaccines during the study.
12. Received any blood products or immunoglobulin products within 3 months prior to enrollment or plan to receive that during the study.
13. Received interferon, systemic corticosteroids, or other immunosuppressants/ immunomodulators (except for local application) for 14 or more consecutive days within 6 months prior to enrollment.
14. Medical history or clinical manifestations of any physical or mental illness that may affect the subject's completion of this study.
15. Needle phobia.
16. Have contraindications for intramuscular administration, such as confirmed thrombocytopenia, any coagulation dysfunction, or being receiving anticoagulation therapy.
17. Have contraindications for electroporation, such as implanted with pacemaker, implanted with Automatic Implantable Cardioverter Defibrillator (AICD), or abnormal electrocardiogram at screening as determined by the investigator.
18. Any other conditions considered by the investigator as not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Frequencies of cross-reactive receptor binding domain (RBD)-specific IFN-γ producing T cells at Day 14 | Day 14
  Frequencies of cross-reactive receptor binding domain (RBD)-specific RBD-specific IFN-γ producing T cells at Day 14 after ICCOV administration compared to baseline (Day 0), as measured by numbers of IFN-γ+ spot-forming unit /1 million PBMC by ELISpot assay.
Frequencies of cross-reactive receptor binding domain (RBD)-specific IFN-γ producing T cells at Day 28 | Day 28
  Frequencies of cross-reactive receptor binding domain (RBD)-specific RBD-specific IFN-γ producing T cells at Day 28 after ICCOV administration compared to baseline (Day 0), as measured by numbers of IFN-γ+ spot-forming unit /1 million PBMC by ELISpot assay.
Frequencies of cross-reactive receptor binding domain (RBD)-specific CD4+ T cells at Day 14 | Day 14
  Frequencies of cross-reactive RBD-specific CD4+ T cell responses at Day 14 after ICCOV administration compared to baseline (Day 0), as analyzed by flow cytometry-based intracellular cytokine staining assays.
Frequencies of cross-reactive receptor binding domain (RBD)-specific CD4+ T cells at Day 28 | Day 28
  Frequencies of cross-reactive RBD-specific CD4+ T cell responses at Day 28 after ICCOV administration compared to baseline (Day 0), as analyzed by flow cytometry-based intracellular cytokine staining assays.
Frequencies of cross-reactive receptor binding domain (RBD)-specific CD8+ T cells at Day 14 | Day 14
  Frequencies of cross-reactive RBD-specific CD8+ T cell responses at Day 14 after ICCOV administration compared to baseline (Day 0), as analyzed by flow cytometry-based intracellular cytokine staining assays.
Frequencies of cross-reactive receptor binding domain (RBD)-specific CD8+ T cells at Day 28 | Day 28
  Frequencies of cross-reactive RBD-specific CD8+ T cell responses at Day 28 after ICCOV administration compared to baseline (Day 0), as analyzed by flow cytometry-based intracellular cytokine staining assays.

SECONDARY OUTCOMES:
Frequencies of cross-reactive receptor binding domain (RBD)-specific IFN-γ producing T cells at Day 60 | Day 60
  Frequencies of cross-reactive receptor binding domain (RBD)-specific RBD-specific IFN-γ producing T cells at Day 60 after ICCOV administration, as measured by numbers of IFN-γ+ spot-forming unit /1 million PBMC by ELISpot assay.
Frequencies of cross-reactive receptor binding domain (RBD)-specific CD8+ T cells at Day 60 | Day 60
  Frequencies of cross-reactive RBD-specific CD8+ T cell responses at Day 60 after ICCOV administration, as analyzed by flow cytometry-based intracellular cytokine staining assays.
Frequencies of cross-reactive receptor binding domain (RBD)-specific CD4+ T cells at Day 60 | Day 60
  Frequencies of cross-reactive RBD-specific CD4+ T cell responses at Day 60 after ICCOV administration, as analyzed by flow cytometry-based intracellular cytokine staining assays.

OTHER OUTCOMES:
Geometric mean titres (GMTs) of neutraliziing antibody against SARS-CoV-2 prototype and epidemic variants | Day 14
  GMTs of neutralizing antibody against SARS-CoV-2 prototype and epidemic variants at Day 14 after ICCOV administration, as measured by pseudovirus-based assay.
Geometric mean titres (GMTs) of neutraliziing antibody against SARS-CoV-2 prototype and epidemic variants | Day 28
  GMTs of neutralizing antibody against SARS-CoV-2 prototype and epidemic variants at Day 28 after ICCOV administration, as measured by pseudovirus-based assay.
Geometric mean titres (GMTs) of neutraliziing antibody against SARS-CoV-2 prototype and epidemic variants | Day 60
  GMTs of neutralizing antibody against SARS-CoV-2 prototype and epidemic variants at Day 60 after ICCOV administration, as measured by pseudovirus-based assay.
Geometric mean increases (GMIs) of neutraliziing antibody against SARS-CoV-2 prototype and epidemic variants | Day 14
  GMIs of neutralizing antibody against SARS-CoV-2 prototype and epidemic variants at Day 14 after ICCOV administration, as measured by pseudovirus-based assay.
Geometric mean increases (GMIs) of neutraliziing antibody against SARS-CoV-2 prototype and epidemic variants | Day 28
  GMIs of neutralizing antibody against SARS-CoV-2 prototype and epidemic variants at Day 28 after ICCOV administration, as measured by pseudovirus-based assay.
Geometric mean increases (GMIs) of neutraliziing antibody against SARS-CoV-2 prototype and epidemic variants | Day 60
  GMIs of neutralizing antibody against SARS-CoV-2 prototype and epidemic variants at Day 60 after ICCOV administration, as measured by pseudovirus-based assay.
Seroconversion rates (SCRs) of neutraliziing antibody against SARS-CoV-2 prototype and epidemic variants | Day 14
  SCRs of neutralizing antibody against SARS-CoV-2 prototype and epidemic variants at Day 14 after ICCOV administration, as measured by pseudovirus-based assay.
Seroconversion rates (SCRs) of neutraliziing antibody against SARS-CoV-2 prototype and epidemic variants | Day 28
  SCRs of neutralizing antibody against SARS-CoV-2 prototype and epidemic variants at Day 28 after ICCOV administration, as measured by pseudovirus-based assay.
Seroconversion rates (SCRs) of neutraliziing antibody against SARS-CoV-2 prototype and epidemic variants | Day 60
  SCRs of neutralizing antibody against SARS-CoV-2 prototype and epidemic variants at Day 60 after ICCOV administration, as measured by pseudovirus-based assay.
Geometric mean titres (GMTs) of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants | Day 14
  GMTs of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants at Day 14 after ICCOV administration, as measured by ELISA.
Geometric mean titres (GMTs) of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants | Day 28
  GMTs of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants at Day 28 after ICCOV administration, as measured by ELISA.
Geometric mean titres (GMTs) of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants | Day 60
  GMTs of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants at Day 60 after ICCOV administration, as measured by ELISA.
Geometric mean increases (GMIs) of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants | Day 14, Day 28, and Day 60
  GMIs of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants at Day 14, 28, and 60 after ICCOV administration, as measured by ELISA.
Geometric mean increases (GMIs) of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants | Day 28
  GMIs of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants at Day 14, 28, and 60 after ICCOV administration, as measured by ELISA.
Geometric mean increases (GMIs) of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants | Day 60
  GMIs of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants at Day 60 after ICCOV administration, as measured by ELISA.
Seroconversion rates (SCRs) of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants | Day 14
  SCRs of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants at Day 14 after ICCOV administration, as measured by ELISA.
Seroconversion rates (SCRs) of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants | Day 28
  SCRs of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants at Day 28 after ICCOV administration, as measured by ELISA.
Seroconversion rates (SCRs) of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants | Day 60
  SCRs of anti-RBD binding antibody against SARS-CoV-2 prototype and epidemic variants at Day 60 after ICCOV administration, as measured by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Fan-ngai, Ivan Hung, Dr., Principal Investigator — The University of Hong Kong
Locations (1):
- Gleneagles Hospital Hong Kong, Wong Chuk Hang, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wong YC, Hang Ho DH, Zhou R, Zhang R, Woo KF, Cheng WY, Wang T, Du Y, Polly Pang KP, Tai WK, Jin X, Chen Z, Ngai Hung IF. An open-label study on the safety and immunogenicity of a PD-1-enhanced DNA vaccine used as a T cell booster for COVID-19. EBioMedicine. 2025 May;115:105699. doi: 10.1016/j.ebiom.2025.105699. Epub 2025 Apr 16. PMID 40245494